CLINICAL TRIAL: NCT03748147
Title: Cervical Ripening in Obese Women: a Prospective, Randomized Trial Comparing Efficacy of 25 mcg Versus 50 mcg of Misoprostol
Brief Title: Cervical Ripening in Obese Women: Efficacy of 25 mcg Versus 50 mcg of Misoprostol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Carri Warshak, Associate Clinical Professor, University of Cincinnati
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016-4435
Record Dates: First submitted 2018-02-22; First posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Induction of Labor Affected Fetus / Newborn
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Intervention Model Description: Parallel design randomized trial. Two study groups: control (25 mcg) intervention (50 mcg)
Who Masked: Participant, Care Provider, Investigator
Masking Description: Both arms will receive identical appearing drug made by the Investigational Drug Unit of the Pharmacy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Standard of care, misoprostol 25 mcg po every four hours
  Interventions: Drug: Misoprostol
- Intervention (Experimental): Misoprostol 50 mcg po every four hours
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — prostaglandin e1
  Other Names: cytotec

SUMMARY:
This is a prospective clinical trial to determine if 50 mcg versus 25 mcg po every four hours of misoprostol has improved efficacy and similar safety in obese women undergoing cesarean section.

DETAILED DESCRIPTION:
We will perform a prospective, randomized, double-blind clinical trial with parallel assignment.

Obese women (delivery BMI 30 or more) who agree to participation will be randomly designated to receive either 25 mcg po q 4 hour (control) misoprosol versus 50 mcg po q 4 hours. Our primary outcome will be the rate of successful induction. Secondary outcomes will include ability to achieve a Bishop score greater than 7, time to active labor, and safety data including rate of tachysystole, non-reassuring fetal status, NICU admission.

ELIGIBILITY:
Inclusion Criteria:

* Labor induction, BMI of 30 or greater, English speaking

Exclusion Criteria:

* Prior cesarean section, uterine tachysystole (5 contractions/ 10 minutes) on admission, Contraindication to labor induction

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnancy, Study of labor induction
Enrollment: 300 (Estimated)
Dates: Start 2018-12-10 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Vaginal delivery | Variable, but within 4 days
  Successful induction defined as a vaginal delivery following labor induction.

SECONDARY OUTCOMES:
Completed cervical ripening | 2 days
  Bishop score of greater than 7 (Bishop score designated per protocol based upon cervical dilation, effacement, station, consistency and position).
Specific time interval from start of induction to active labor | 2 days
  We will measure the interval (hours) between start of cervical ripening and active labor defined as reaching a cervical dilation of 6 cm.
Rate of tachysystole, fetal nonreassuring status, uterine rupture | 3 days
  Rate of the following as categorical variables: tachysystole (any delay in study medication administration for greater than 5 contractions/10 minute window), non-reassuring fetal status (any evaluation of the fetal tracing that leads to delays in study drug administration secondary to concerns for the fetal status), NICU admission, uterine rupture

IPD SHARING:
Plan to Share IPD: Undecided
Would consider upon request.